CLINICAL TRIAL: NCT01710644
Title: A Randomized, Double-blind, Multicenter, Two-period Crossover Study to Assess the Efficacy and Tolerability of NM-BL (Burlulipase) in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Brief Title: Efficacy and Tolerability of NM-BL in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nordmark Arzneimittel GmbH & Co. KG (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM-BL-101; 207862 (Other: Parexel)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Pancreatic Insufficiency; Cystic Fibrosis; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis; Digestive System Diseases; Lung Diseases; Respiratory Tract Diseases | interventions — caramel coloring

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Burlulipase (Experimental): Burlulipase orally, per meal
  Interventions: Drug: Burlulipase
- Placebo (Caramel in sterile water) (Placebo Comparator): Placebo orally, per meal
  Interventions: Drug: Placebo (Caramel in sterile water)

INTERVENTIONS:
Drug: Burlulipase — Burlulipase oral solution will be taken with meals and snacks for 5 to 7 days
  Other Names: NM-BL
  Arms: Burlulipase
Drug: Placebo (Caramel in sterile water) — Placebo will be taken with meals and snacks for 5 to 7 days
  Other Names: Placebo
  Arms: Placebo (Caramel in sterile water)

SUMMARY:
The purpose of this Randomized, Double-blind, Multicenter, Two-period Crossover Study is to Assess the Efficacy and Tolerability of Burlulipase (NM-BL) in Patients with Exocrine Pancreatic Insufficiency due to Cystic Fibrosis

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥12 years from the date of informed consent
* Confirmed diagnosis of CF at screening
* Confirmed EPI by historical (within past 12 months) CFA <70% without use of PERTs or current fecal elastase <50 µg/g stool at screening
* Currently receiving PERT with a commercially available pancreatic enzyme
* Currently on stable treatment with proton pump inhibitors or H2 receptor antagonists
* Clinically stable condition without evidence of acute respiratory disease or any other acute condition

Exclusion Criteria:

* History of fibrosing colonopathy
* History of significant bowel resection, in the opinion of the investigator, or solid organ transplant
* History of being refractory to pancreatic enzyme replacement
* Current diagnosis or history of distal intestinal obstruction syndrome
* Current diagnosis of small intestinal bacterial overgrowth, ileus or acute abdomen
* A body mass index percentile <10%

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of NM-BL compared to placebo in patients with Exocrine Pancreatic Insufficiency (EPI) due to CF, where the primary variable is coefficient of fat absorption (CFA%) | 72 hrs

SECONDARY OUTCOMES:
To evaluate the efficacy of NM-BL compared to placebo in patients with Exocrine Pancreatic Insufficiency (EPI)due to CF, where the primary variable is coefficient of nitrogen absorption (CNA%) | 72 hrs

OTHER OUTCOMES:
Symptomatology / Symptom Questionnaire | 7 days
  Comparison gastrointestinal parameters, recorded by the patient/carer in the Symptom Questionnaire each day during the Treatment Periods

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Forssmann, MD, Study Director — Nordmark Arzneimittel GmbH & Co. KG; James E. Heubi, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (9):
- United States (9):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - The University of Iowa, Iowa City, Iowa
  - Via Cristi Hospitals Wichita, Inc., Wichita, Kansas
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - West Virginia University Research Corporation, Morgantown, West Virginia

REFERENCES:
- [Derived] Somaraju URR, Solis-Moya A. Pancreatic enzyme replacement therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Aug 5;8(8):CD008227. doi: 10.1002/14651858.CD008227.pub4. PMID 32761612
- [Derived] Heubi JE, Schaeffer D, Ahrens RC, Sollo N, Strausbaugh S, Graff G, Jain R, Witte S, Forssmann K. Safety and Efficacy of a Novel Microbial Lipase in Patients with Exocrine Pancreatic Insufficiency due to Cystic Fibrosis: A Randomized Controlled Clinical Trial. J Pediatr. 2016 Sep;176:156-161.e1. doi: 10.1016/j.jpeds.2016.05.049. Epub 2016 Jun 11. PMID 27297209